CLINICAL TRIAL: NCT02904239
Title: Evaluation of Cardiac Pathologies in Standard Thoracic CT Imaging [CaPaCT]
Brief Title: Cardiac Pathologies in Standard Thoracic CT Imaging
Acronym: CaPaCT
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-4-116
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease
Keywords: Multidetector Computed Tomography; Incidental cardiac findings; Thoracic high-pitch Computed Tomography; Management guidelines
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Modern high-end CT scanners with faster scan acquisition times now allow for routine assessment of cardiac pathologies, which could result in numerous incidental cardiac findings on standard thoracic CT angiography (CTA) scans. The CaPaCT-study aims to assesses the presence, management and possible clinical impact of incidental cardiac pathologies which are becoming visible on standard thoracic CT scans performed on new high-end scanners.

DETAILED DESCRIPTION:
A known disadvantage of constantly improving diagnostic imaging is the detection of incidental findings. Computed Tomography (CT) scanner technology is ever improving in both temporal and spatial resolution. Recently developed advanced reconstruction algorithms and dedicated post-processing software reduce image noise thereby improving image quality. Equipped with these advancements, modern CT scanners accomplish well defined imaging of cardiovascular structures. These technical improvements have enabled cardiac assessment on routine standard (non-ECG triggered) thoracic CT scans.

If thoracic radiologists are able to assess the heart and coronary arteries on a standard thoracic CT, this could result in an extensive amount of incidental cardiac findings. Herein lies the potential for large scale reporting of incidental cardiac findings and, consequently, a huge influx of new 'patients' for downstream testing and potential (over-)treatment.

Coronary Artery Disease (CAD) is a known comorbidity for multiple diseases, for example presence of CAD could require a different treatment strategy in lung cancer and worsen prognosis [Khakoo et al]. In patients with diabetes mellitus (DM), the incidence of CAD is four times higher compared with the general population, and the risk of a cardiovascular event is two- to four-fold higher [Kannel et al. + Aktas et al.]. Therefore, the discussion on management and treatment of these patients with incidental cardiac findings on chest CT evidently is important. Unfortunately, to date no consensus has been reached on the management and reporting of these findings. The CaPaCT study (cardiac pathologies on standard thoracic CT) has been developed to evaluate the visibility and management of incidental cardiac pathologies on a ultra-high pitch thoracic CT-scan with help of the CAD-RADS classification.

ELIGIBILITY:
Inclusion Criteria:

- Standard non-ECG triggered thoracic CT scanning.

Exclusion Criteria:

* Iodine allergy
* Renal insufficiency (GFR < 30mL/min)
* Pregnancy
* Age < 18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients referred for thoracic CT-scanning.
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2016-07; Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Evaluate visibility and management of coronary artery disease (CAD) | One year
  Evaluating visibility and management of CAD on standard thoracic CT with help of the CAD-RAD system.

SECONDARY OUTCOMES:
Objective image quality | One year
  Objective image quality of standard thoracic CT scans
Subjective image quality | One year
  Subjective image quality of standard thoracic CT scans

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khakoo AY, Yeh ET. Therapy insight: Management of cardiovascular disease in patients with cancer and cardiac complications of cancer therapy. Nat Clin Pract Oncol. 2008 Nov;5(11):655-67. doi: 10.1038/ncponc1225. Epub 2008 Sep 16. PMID 18797437
- [Background] Kannel WB, McGee DL. Diabetes and cardiovascular disease. The Framingham study. JAMA. 1979 May 11;241(19):2035-8. doi: 10.1001/jama.241.19.2035. PMID 430798
- [Background] Aktas MK, Ozduran V, Pothier CE, Lang R, Lauer MS. Global risk scores and exercise testing for predicting all-cause mortality in a preventive medicine program. JAMA. 2004 Sep 22;292(12):1462-8. doi: 10.1001/jama.292.12.1462. PMID 15383517